CLINICAL TRIAL: NCT02647658
Title: Targeted Interventions to Prevent Chronic Low Back Pain in High Risk Patients: A Multi-Site Pragmatic Cluster Randomized Controlled Trial
Brief Title: Targeted Interventions to Prevent Chronic Low Back Pain in High Risk Patients
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Boston Medical Center (Other); Intermountain Health Care, Inc. (Other); Johns Hopkins University (Other); Medical University of South Carolina (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Anthony Delitto, Professor and Dean, SHRS, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS-1402-10867
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
Keywords: acute low back pain; primary care; psychologically informed physical therapy; cluster randomized pragmatic trial; comparative effectiveness; secondary prevention
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Parallel assignment of clusters (clinics). Cluster randomized trial.
Oversight: Data Monitoring Committee: No

ARMS (2):
- GBC+PIPT (Experimental): Guideline Based Care plus Psychologically Informed Physical Therapy (GBC+PIPT)
  Interventions: Behavioral: Guideline Based Care plus Psychologically Informed Physical Therapy
- GBC (Active Comparator): Guideline Based Care (GBC)
  Interventions: Behavioral: Guideline Based Care (GBC)

INTERVENTIONS:
Behavioral: Guideline Based Care plus Psychologically Informed Physical Therapy — PCP care is enhanced with a prompt referral to physical therapy (PT) that includes psychologically informed coaching directed towards education and reduced fear of movement
  Arms: GBC+PIPT
Behavioral: Guideline Based Care (GBC) — Management decisions are made between PCPs and patients with the guidance of best evidence but with no specific directives
  Arms: GBC

SUMMARY:
Low back pain (LBP) is a common problem among US adults. Initial episodes tend to be self-limited ("acute"), but some people can progress to a state of persistent pain. Often termed "chronic" LBP (cLBP), this condition can cause prolonged difficulty with most daily activities, including job performance. This study will compare two approaches for preventing patients with acute LBP (aLBP) from developing cLBP using a pragmatic, cluster randomized trial. The first approach is to provide PCPs with information regarding a patient's risk of transitioning from aLBP to cLBP and to encourage PCPs to treat patients according to accepted clinical guidelines. The second approach is to provide the same risk information and have PCPs team up with physical therapists to deliver psychologically-informed physical therapy (PIPT) for those patients determined to be at high risk for transitioning to cLBP. The 1,860 patients expected to be enrolled at five regional sites (Pittsburgh, Pennsylvania; Boston, Massachusetts; Baltimore, Maryland; Charleston, South Carolina; and Salt Lake City, Utah) will start the study when their LBP is in an acute phase. The study's primary aims are to compare the proportions of cLBP and measures of functional ability between the two groups at 6 months. Secondary aims are to measure the referrals to physical therapists and specialists, opioid prescriptions, LBP-related x-rays or MRIs, surgeries, and other medical procedures during a 12-month follow-up period.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common problem among US adults. Initial episodes tend to be self-limited ("acute"), but some people can progress to a state of persistent pain. Often termed "chronic" LBP (cLBP), this condition can cause prolonged difficulty with most daily activities, including job performance. Most patients see chiropractors or primary care physicians (PCPs) for initial episodes of LBP. This study will compare two approaches for preventing patients with acute LBP (aLBP) from developing cLBP using a cluster randomized trial. Both treatments can be delivered in an outpatient PCP setting. The first approach is to provide PCPs with information regarding a patient's risk of transitioning from aLBP to cLBP and to encourage PCPs to treat patients according to accepted clinical guidelines (Guideline Based Care, GBC). The second approach is to provide the same risk information and have PCPs team up with physical therapists to deliver psychologically-informed physical therapy (PIPT) for those patients determined to be at high risk for transitioning to cLBP (GBC+PIPT). PIPT is designed to help patients identify and overcome physical and psychological barriers to recovery. The 1,860 patients expected to be enrolled as part of quality improvement at five regional sites (Pittsburgh, Pennsylvania; Boston, Massachusetts; Baltimore, Maryland; Charleston, South Carolina; and Salt Lake City, Utah) will start the study when their LBP is in an acute phase. The study's primary aims are to compare the proportions of cLBP and measures of functional ability between the two groups at 6 months. Secondary aims are to measure the referrals to physical therapists and specialists, opioid prescriptions, LBP-related x-rays or MRIs, surgeries, and other medical procedures during a 12-month follow-up period. This study was designed with input from a variety of national and local stakeholders, including patients with LBP, providers, payers, professional organizations, purchasers, and policy representatives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Receiving care for acute low back pain during a primary care clinic visit
* Able to provide informed consent

Exclusion Criteria:

* Medical contraindications to physical therapy based on the judgment of the primary care provider as documented in the medical record (i.e., "red flag" signs and symptoms of a potentially serious condition such as cauda equina syndrome, major or rapidly progressing neurological deficit, cancer, spinal infection or fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Delitto, PT, PhD, Principal Investigator — University of Pittsburgh; Robert Saper, MD, MPH, Principal Investigator — Boston Medical Center
Locations (5):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Intermountain Healthcare, Salt Lake City, Utah

REFERENCES:
- [Derived] Roseen EJ, Smith CN, Essien UR, Cozier YC, Joyce C, Morone NE, Phillips RS, Gergen Barnett K, Patterson CG, Wegener ST, Brennan GP, Delitto A, Saper RB, Beneciuk JM, Stevans JM. Racial and Ethnic Disparities in the Incidence of High-Impact Chronic Pain Among Primary Care Patients with Acute Low Back Pain: A Cohort Study. Pain Med. 2023 Jun 1;24(6):633-643. doi: 10.1093/pm/pnac193. PMID 36534910
- [Derived] Beneciuk JM, George SZ, Patterson CG, Smith CN, Brennan GP, Wegener ST, Roseen EJ, Saper RB, Delitto A. Treatment effect modifiers for individuals with acute low back pain: secondary analysis of the TARGET trial. Pain. 2023 Jan 1;164(1):171-179. doi: 10.1097/j.pain.0000000000002679. Epub 2022 May 9. PMID 35543647
- [Derived] Delitto A, Patterson CG, Stevans JM, Freburger JK, Khoja SS, Schneider MJ, Greco CM, Freel JA, Sowa GA, Wasan AD, Brennan GP, Hunter SJ, Minick KI, Wegener ST, Ephraim PL, Beneciuk JM, George SZ, Saper RB. Stratified care to prevent chronic low back pain in high-risk patients: The TARGET trial. A multi-site pragmatic cluster randomized trial. EClinicalMedicine. 2021 Mar 30;34:100795. doi: 10.1016/j.eclinm.2021.100795. eCollection 2021 Apr. PMID 33870150
- [Derived] Middleton A, Fitzgerald GK, Delitto A, Saper RB, Gergen Barnett K, Stevans J. Implementing stratified care for acute low back pain in primary care using the STarT Back instrument: a process evaluation within the context of a large pragmatic cluster randomized trial. BMC Musculoskelet Disord. 2020 Nov 25;21(1):776. doi: 10.1186/s12891-020-03800-6. PMID 33238964
- [Derived] Delitto A, Patterson CG, Stevans JM, Brennan GP, Wegener ST, Morrisette DC, Beneciuk JM, Freel JA, Minick KI, Hunter SJ, Ephraim PL, Friedman M, Simpson KN, George SZ, Daley KN, Albert MC, Tamasy M, Cash J, Lake DS, Freburger JK, Greco CM, Hough LJ, Jeong JH, Khoja SS, Schneider MJ, Sowa GA, Spigle WA, Wasan AD, Adams WG, Lemaster CM, Mishuris RG, Plumb DL, Williams CT, Saper RB. Study protocol for targeted interventions to prevent chronic low back pain in high-risk patients: A multi-site pragmatic cluster randomized controlled trial (TARGET Trial). Contemp Clin Trials. 2019 Jul;82:66-76. doi: 10.1016/j.cct.2019.05.010. Epub 2019 May 25. PMID 31136834
- [Derived] Beneciuk JM, George SZ, Greco CM, Schneider MJ, Wegener ST, Saper RB, Delitto A. Targeted interventions to prevent transitioning from acute to chronic low back pain in high-risk patients: development and delivery of a pragmatic training course of psychologically informed physical therapy for the TARGET trial. Trials. 2019 May 6;20(1):256. doi: 10.1186/s13063-019-3350-3. PMID 31060589

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Primary Care Clinics
Groups:
- Guideline Based Care: Guideline Based Care (GBC)
  Guideline Based Care (GBC): Management decisions are made between PCPs and patients with the guidance of best evidence but with no specific directives
Period: Overall Study
Arm/Group | GBC+PIPT | Guideline Based Care
Started | 1207; 39 Primary Care Clinics | 1093; 37 Primary Care Clinics
6 Month Assessment | 658; 38 Primary Care Clinics | 635; 35 Primary Care Clinics
Completed | 1192; 39 Primary Care Clinics | 1069; 37 Primary Care Clinics
Not Completed | 15; 0 Primary Care Clinics | 24; 0 Primary Care Clinics
Not completed — Consent refusal | 15 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GBC+PIPT | Guideline Based Care | Total
Number analyzed (Participants) | 1207 | 1093 | 2300
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (16.2) | 50.6 (17.1) | 49.9 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 721 | 635 | 1356
  Male | 486 | 458 | 944
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 72 | 147
  Not Hispanic or Latino | 1087 | 995 | 2082
  Unknown or Not Reported | 45 | 26 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race from electronic medical record
  Participants
    Race: White | 949 | 769 | 1718
    Race: Black | 181 | 224 | 405
    Race: Other | 25 | 57 | 82
    Race: Missing/Unknown | 52 | 43 | 95
Oswestry Disability Index [Mean (Standard Deviation); unit: score on scale] — Oswestry Low Back Pain Disability Questionnaire. A measure of a patient's functional disability. The scale ranges from 0% to 100% with higher scores indicating more disability. Population: All of those patients who completed the survey.
  score on scale
    number analyzed (Participants) | 1161 | 1063 | 2224
    (all) | 48.0 (17.4) | 48.3 (17.5) | 48.1 (17.4)
STarT Back Total [Mean (Standard Deviation); unit: score on a scale] — STarT Back Screening Tool for Risk Stratification, ranges from 0 to 9 with higher scores indicating higher risk for persistent disabling symptoms. It is designed to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making.
  score on a scale | 7.2 (1.1) | 7.2 (1.1) | 7.2 (1.1)
STarT Back Subscore [Mean (Standard Deviation); unit: score on a scale] — Questions 5 to 9 of the STarT Back Screening Tool for Risk Stratification. The distress subscale score is used to identify the high-risk subgroup. The items are fear, anxiety, catastrophising, depression and bothersomeness. Subscale scores range from 0 to 5 with patients scoring 4 or 5 being classified into the high-risk subgroup
  score on a scale | 4.4 (0.5) | 4.3 (0.5) | 4.4 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Reported Transition From Acute to Chronic Low Back Pain (cLBP)
Description: Measured using a 2-item Chronic Low Back Pain (LBP) questionnaire. Patient endorses low back pain that interferes with regular daily activities more than 3 months and more then 1/2 the days in the past 6 months.
Time Frame: 6 months from baseline
Population: Among participants with assessment data at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 658 | 635
Participants | 312 | 318

2. Primary Outcome: Functional Disability
Description: Measured using the 10-item Oswestry Disability Index (version 2.1a). Also known as the Oswestry Low Back Pain Disability Questionnaire.
  A measure of a patient's functional disability. The scale ranges from 0% to 100% with higher scores indicating more disability.
Time Frame: 6 months
Population: Participants with assessment data at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 658 | 635
score on a scale | 27.3 [25.4 to 29.3] | 29.5 [27.5 to 31.5]

3. Secondary Outcome: Number of Patients Referred to Physical Therapy
Description: Patient referred to physical therapy or psychologically informed physical therapy measured using electronic health records over 12 months.
Time Frame: 12 months
Population: All screened excluding those not consented for EMR follow up at 12 months at 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 106 | 77

4. Secondary Outcome: Number of Patients Prescribed Opioids
Description: Medication prescription for opioids measured using electronic health records over 12 months.
Time Frame: 12 months
Population: All screened excluding patients that did not consent to EMR data at 12 months at 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 89 | 86

5. Secondary Outcome: Number of Patients With Orders for Diagnostic Imaging Tests
Description: Referrals for diagnostic imaging (X-rays and MRI) measured using electronic health records
Time Frame: 12 months
Population: All screened except participants who did not provide consent for 12 month follow up from EMR from 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 74 | 73

6. Secondary Outcome: Number of Patients Referred to Other Rehabilitation or Pain Management Specialist
Description: Referral to any non-physical therapy rehabilitation or pain management specialist (chiropractic, physiatrist, pain management) measured using electronic health records
Time Frame: 12 months
Population: All screened except participants who did not provide consent for 12 month follow up from EMR from 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 45 | 26

7. Secondary Outcome: Number of Patients Referred to Surgery Specialist
Description: Referral to any surgical specialist (orthopaedist, neurosurgeon, anesthesiologist) measured using electronic health records
Time Frame: 12 months
Population: All screened except participants who did not provide consent for 12 month follow up from EMR from 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 38 | 44

8. Secondary Outcome: Number of Patients Undergoing Interventional Pain Procedures
Description: Receipt of interventional pain procedures including epidural steroid injections measured using electronic health records
Time Frame: 12 months
Population: All screened except participants who did not provide consent for 12 month follow up from EMR from 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 32 | 43

9. Secondary Outcome: Number of Patients Who Had Back Surgery
Description: Documentation that patient underwent back surgery in electronic health records
Time Frame: 12 months
Population: All screened except participants who did not provide consent for 12 month follow up from EMR from 1 site.
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1192 | 1069
Participants | 29 | 19

10. Other Pre Specified Outcome: Number of Patients Prescribed Opioids
Description: Medication prescription for opioids measured using electronic health records at the index baseline visit for the patient. Measure of intervention fidelity post clinic randomization.
Time Frame: Up to 21 days after initial visit for acute low back pain
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1207 | 1093
Participants | 300 | 270

11. Other Pre Specified Outcome: Number of Patients Referred to Physical Therapy
Description: Patient referred to physical therapy or psychologically informed physical therapy measured using electronic health records at the index baseline visit. This is a measure of intervention fidelity post-randomization of the clinics.
Time Frame: Up to 21 days after initial visit for acute low back pain
Measure: Count of Participants; unit: Participants
Arm/Group | GBC+PIPT | Guideline Based Care
Number analyzed (Participants) | 1207 | 1093
Participants | 658 | 335

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: The TARGET trial was a pragmatic trial in four health care systems. As such, we did not collect data on adverse events.
Arm/Group | GBC+PIPT | Guideline Based Care
All-Cause Mortality (participants affected / at risk) | 8/1207 | 12/1093
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT02647658/Prot_SAP_000.pdf